CLINICAL TRIAL: NCT03277768
Title: Non-Invasive Detection of Tissue Oxygen Deprivation in Premature Infants With Patent Ductus Arteriosus.
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201601508
Record Dates: First submitted 2017-09-01; First posted 2017-09-11 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Premature Infant; Patent Ductus Arteriosus; Hemodynamic Instability
Keywords: Premature infant; Tissue Oxygenation; Patent Ductus Arteriosus
MeSH Terms: conditions — Premature Birth; Ductus Arteriosus, Patent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group -Patent Ductus Arteriosus Absent
  Interventions: Device: Resonance Raman Spectroscopy (RRS)
- Study Group - Patent Ductus Arteriosus Present
  Interventions: Device: Resonance Raman Spectroscopy (RRS)

INTERVENTIONS:
Device: Resonance Raman Spectroscopy (RRS) — Pre and post-ductal RRS measurements will be obtained daily for a maximum of 14 data collection times in infants with and without PDAs.

SUMMARY:
The proposed research evaluates tissue oxygenation (StO2) as measured by resonance raman spectroscopy (RRS) in premature infants with and without patent ductus arteriosus (PDA). This is a prospective observational study of infants born at < 30 weeks of gestation. The primary aim of this study is to determine if the difference in pre- and post-ductal StO2 as detected by RRS is more significant in premature infants with PDA in comparison to infants without PDA. The secondary aim of this study is to determine if the difference in pre- and post-ductal StO2 as detected by RRS is more significant in infant who develop serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Infants < 30 weeks estimated gestational age

Exclusion Criteria:

* Infants with major congenital anomalies
* Infants >34 weeks post-menstrual age

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Premature infants born <30 weeks gestational age and admitted to the Boston Children's Hospital neonatal intensive care unit (NICU), Brigham and Women's NICU, and the University of Florida NICU.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-08-23 (Actual)

PRIMARY OUTCOMES:
Differences and pre- and post-ductal RRS measurements of tissue oxygenation. | Up to a maximum of 14 data collection times
  Pre- and post-ductal tissues oxygenation as measured by RRS may be more significant in infants with PDA.

SECONDARY OUTCOMES:
Are differences in pre- and post-ductal StO2 as detected by RRS more significant in infants with serious adverse events. | Up to a maximum of 14 data collection times
  RRS measurements and the difference between pre- and post-ductal tissue oxygenation will be evaluated in infants with serious adverse events to determine if the measurements could have predicted the serious adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: J Lauren Ruoss, MD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - Boston Children's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No
The analysis of the data will be shared with other research. Individual patient data will not be shared.